CLINICAL TRIAL: NCT01043016
Title: Safety Study of Photodynamic Therapy Using Photocyanine Injection in Treating Patients With Malignant Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Longhua Pharmaceutical Co. Ltd (Other)
Collaborators: Fuzhou University (Other); Sun Yat-sen University (Other)
Responsible Party: Safety Study of Photodynamic Therapy Using Photocyanine Injection in Treating Patients With Malignant Tumors, Fujian Longhua Pharmaceutical Co. Ltd
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008L03278
Record Dates: First submitted 2010-01-04; First posted 2010-01-06 (Estimated); Last update posted 2010-01-06 (Estimated); Status verified 2010-01

CONDITIONS: Skin Cancer; Esophageal Cancer
Keywords: skin cancer; esophageal cancer; photodynamic therapy
MeSH Terms: conditions — Skin Neoplasms; Esophageal Neoplasms | interventions — Photochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Photocyanine injection (Experimental): Patients receive intravenous injection of Photocyanine injection from dosage of 0.1 mg/kg,0.2 mg/kg,0.33 mg/kg,0.5 mg/kg to 0.6 6mg/kg till the dose-limiting effect occur.
  Interventions: Procedure: Photodynamic therapy

INTERVENTIONS:
Procedure: Photodynamic therapy — patient undergo Photocyanine Injection via venous infusion followed by photodynamic therapy with 670nm diobe laser 24 hours later

SUMMARY:
The purpose of this study is to determine the safety and maximum tolerated dose of Photocyanine injection in photodynamic therapy of malignant tumor (especially skin cancer and esophageal cancer).

Projected accrual: A total of 18-24 patients will be accrued for this study.

DETAILED DESCRIPTION:
Photocyanine injection is a type of cyanine compound, which was invented in Fuzhou university by Professor Chen; it's maximum absorption wave is 670 nm. Patients receive intravenous injection of Photocyanine injection, and 24 hours later, patients undergo photodynamic therapy.

Cohorts of 3-6 patients receive escalating doses of Photocyanine Injection and photodynamic therapy until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 1 of 3 patients experiences dose-limiting toxicity. Three additional patients are treated at the MTD.

After completion of study therapy, patients are followed for up to 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 70 years old (patient over 60 years old must not have three kinds of complications of heart, lung, liver and kidney function at the same time), no gender limited;
2. Advanced malignant solid tumors confirmed by histology or cytology ( skin cancer and esophageal cancer), malignant tumor can be illuminated directly (or via endoscopy) by the laser fiber;
3. Recurrence after surgery, radiotherapy,chemoradiotherapy; or have financial difficulties, give up any other treatment;
4. Patients received chemotherapy, biological therapy or other research drugs must exceed at least 4 weeks or more than five half-life;
5. Life expectancy: > 3 months;
6. Can collaboratively observe the adverse events and efficacy;
7. No other anti-tumor treatment (including steroids);
8. Patients or their legal representative can sign the informed consent;
9. Performance status: ECOG ≤ 2,

Exclusion Criteria:

1. No pathological evidence;
2. Have allergic effect to this drug;
3. HIV antibody positive, or suffering from other acquired and congenital immune deficiency diseases, or have organ transplant history;
4. Neutrophil count < 1.5 × 109 / L, platelet < 100 × 109 / L, or hemoglobin < 90 g /L;
5. Serum Cr above 1.5 times of normal reference range or Cr clearance rate < 50 ml/min;
6. ALT, or AST > 2.5 times of the normal range when no hepatic metastasis occur; or ALT, or AST > 5 times of the normal range when hepatic metastasis exist;
7. Serum bilirubin > 1.5 times of the normal range;
8. Fever above 38 ℃, or have active infection which can affect the clinical trials obviously;
9. Hypertension failed to be controlled (systolic blood pressure > 160 mmHg or diastolic pressure > 100 mmHg);
10. Obvious cardiovascular disorders (eg, myocardial infarction, superior vena cava syndrome, more than two grades heart disease, or heart disease which can increase the risk of ventricular arrhythm);
11. Not recover from any anticancer therapy or surgery;
12. Any clinical problems beyond control (such as severe mental, neurological, cardiovascular, respiratory system diseases, etc.);
13. Evidence of central nerve system metastasis;
14. Have some gastrointestinal disease which can affect the distribution, metabolism or removal of this drug;
15. Pregnant or breast-feeding women;
16. Poor compliance.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-03 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | one month

SECONDARY OUTCOMES:
Treatment efficacy as measured by computed tomography (CT) or magnetic resonance imaging (MRI) and endoscopy exam 3 weeks after the start of study treatment according to the Response Evaluation Criteria In Solid Tumors (RECIST) standard | six weeks

CONTACTS AND LOCATIONS:
Overall Officials: guo l xu, Principal Investigator — Sun Yat-sen University
Locations (1):
- Department of Endoscopy and Laser,Sun Yat-Sen University,Cancer Center, Guangzhou, Guangdong, China